CLINICAL TRIAL: NCT02884050
Title: Physiologic Effects of Topiramate on Cognition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 96-2009
Record Dates: First submitted 2016-08-23; First posted 2016-08-30 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Alteration of Cognitive Function
MeSH Terms: interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topiramate (Experimental): single, 100mg oral dose of topiramate
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): matched inactive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — antiepilepsy drug
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo — non-active placebo
  Arms: Placebo

SUMMARY:
Data generated from this pilot project will be used to support a larger, NIH funded study to investigate the physiologic mechanisms associated with the cognitive side effects of a commonly prescribed antiepileptic drug (AED), topiramate (TPM). This study will provide pilot data to 1) demonstrate the viability of using quantitative electroencephalogram (EEG) to examining physiological effects of AEDs as they relate to language function, and 2) perform formal power estimate calculations in support of a longer-term connectivity study using stochastic modeling techniques including power, coherence, and Granger causality metrics to analyze AED effects on quantitative EEG. Traditionally, the cognitive side effects of AEDs have been considered a byproduct of decreased neuronal excitation associated with medical therapy, although recent data suggests that this may not be true for some newer medications, such as TPM. The proposed experiments will employ quantitative EEG to investigate the effects of topiramate on neuronal network connectivity and pharmacokinetic/pharmacogenetic relationships in order to explore individual physiological responses. Topiramate is selected because of its relatively unique effects on generative verbal fluency, but unlike older AEDs, TPM is associated with little EEG change. The investigators will compare the effects of TPM to baseline and an inactive placebo in a randomized double blind crossover design.

DETAILED DESCRIPTION:
Background:

Cognitive side-effects of antiepileptic drugs (AEDs) are important components of treatment tolerability, although the physiologic mechanisms associated with their cognitive effects are poorly understood. Quantitative EEG and other neurophysiologic measures are sensitive indicators of central AED effects and in the older AEDs, with slowing consistent with a diffuse encephalopathy, tend to covary with neuropsychological performance. EEG changes are generally more sensitive than neuropsychological testing to AEDs, and have been demonstrated for oxcarbazepine, phenytoin, carbamazepine, lamotrigine, and levetiracetam.

Recent evidence demonstrates that the cognitive effects of these agents cannot be explained simply by diffuse reduction of neuronal excitability. Older AEDs are associated with a mild-to-moderate generalized cognitive effect such as decreased psychomotor speed, which is also accompanied by encephalopathic EEG patterns including increased spectral EEG power in the lower frequency bands. Several of the newer AEDs have not demonstrated this pattern. Some of these have reduced cognitive effects; however, one of the new AEDs, topiramate (TPM), which also does not possess this EEG encephalopathic pattern, actually produces greater cognitive deficits than many older AEDs.

Although newer AEDs tend to have a more favorable cognitive profile, TPM, which is indicated for partial or primary generalized epilepsy as well as migraine prophylaxis, is being increasingly prescribed for a wide range of neuropsychiatric disorders including bipolar disorder, weight loss and even eating disorders despite carrying a high risk of neuropsychological impairment with a prominent effect on verbal fluency. Although TPM's effect on verbal fluency may reflect a more widespread disruption of frontal lobe function, TPM's effect on verbal fluency has also been interpreted by some as reflecting a more general effect on language. TPM has multiple mechanisms of actions including modification of Na+ or Ca2+ dependent action potentials, enhancement of gamma-aminobutyric acid (GABA)-mediated receptors, and inhibition of kainate-mediated conductance at glutamate receptors of the alpha-amino-3-hydroxy-5-methyl-4-isoxazoleproprionic acid (AMPA)/kainate type. In addition, TPM is a carbonic anhydrase (CA) II inhibitor, and although the functions of CA in the central nervous system (CNS) is not well-established, at least some CA isoenzymes (CA II) have heavy human brain concentrations in oligodendrocytes and myelin. Because TPM is unique in that its neuropsychological effects are not accompanied by quantitative spectral EEG components, a generalized reduction in neuronal excitation is insufficient to account for TPM's neuropsychological profile. Therefore, investigators are investigating whether the physiologic mechanisms underlying TPM's negative cognitive effect is reflected by altered patterns of neuronal EEG connectivity following a single dosing.

TPM's inhibitory effect on carbonic anhydrase suggests that its mechanism of cognitive impairment may be related to white matter dysfunction altering neuronal connectivity. If true, then TPM's effects should be greater on generative fluency than semantic-decision due to disruption of intentional system connectivity of the frontal lobe and anterior cingulate with other brain regions. Semantic-conceptual processing with semantic-decision should be unaffected. However, TPM has multiple mechanisms which may contribute to its cognitive effects. If a generalized "frontal lobe" effect is present, then similar TPM effects should be present for working memory activations. EEG provides the opportunity to explore differential changes in functional connectivity associated with AEDs as a function of task.

In addition, TPM appears to have a significant and selective effect on word finding and verbal fluency in a minority of patients that isn't manifest by other AEDs. As Goldstein et al point out in their recent review, this type of heterogeneity of response may be part be explained by genes involved in both the metabolism and central response to TPM.

The investigators hypothesize that the physiological effects of TPM on cognition are manifest at the functional network level, with the greatest reduction in connectivity expected during verbal fluency. The primary objective of this project is to characterize TPM's effects on working memory and verbal fluency during quantitative EEG recording in healthy volunteers. This study will provide pilot data to 1) demonstrate the viability of this approach to examining physiological effects of AEDs as they relate to language function, and 2) perform formal power estimate calculations in support of a longer-term connectivity study using stochastic modeling techniques including power, coherence, and Granger causality metrics to analyze AED effects on quantitative EEG.

The primary research goal of this project is to establish the relationship of single dose TPM on quantitative cognitive EEG in order to investigate the physiological mechanisms underlying the cognitive effects of AEDs. Investigators will examine neuronal network connectivity and potential pharmacokinetic relationships to individual physiological responses.

Specific Aim 1a. To determine the change in functional EEG connectivity following single dose TPM compared to placebo during a working memory task.

The secondary research goal of this project is to collect preliminary data on the genetics of TPM metabolism and genetic influences on TPM-induced changes in verbal fluency and working memory.

Specific Aim 2. To investigate the association between genotype and changes in verbal fluency and working memory as a result of taking a single 100 mg TPM versus a placebo.

Design: This is a double-blind, placebo-controlled, double crossover study designed to investigate the physiologic effect of a single dose of TPM (100 mg) or placebo on cognition and working memory. Subjects will undergo cognitive EEG recording, neuropsychological testing and blood draws.

Informed Consent:

The nature of the research study and the possible risks will be explained to each potential subject. The subjects will be made aware that their medical care is not contingent on their participation. Written informed consent will be obtained from each subject by one of the co-investigators.

Design Overview:

On the study days, subjects will be initially directed to the University of Florida (UF)

Neuroinformatics Lab in the J. Crayton Pruitt Family Department of Biomedical Engineering:

* After signing the informed consent, subjects will be randomly assigned to a study treatment sequence. All medication will be purchased by the UF Pharmacy. Subjects will be asked to abstain from alcoholic beverages or over-the-counter medications for at least 48 hours prior to testing though they will be permitted to consume caffeinated beverages on the day of their assessment if that is part of their standard morning routine.
* After being ask to consent to the study, a brief demographic, medical and medication history will be taken on the first visit to assure that subjects are not currently on any medications that can interact with either TPM.
* Vital signs will be recorded.
* Subject will be fitted with EEG electrodes. On the 2nd and 3rd visits, study medication will be consumed just prior to the electrode placement.
* After completing the EEG recording session (approx. 2.5 hours), electrodes will be removed, Blood will be drawn for serum concentrations (a genetic sample will be taken at this time on the first visit ONLY after separate consent is obtained).
* The subject will then be given a small snack after which a brief neuropsychological assessment (~ 20 minutes) will be administered by a blinded tester.

This same procedure will be repeated at least one week apart until all study conditions have been obtained. All testing will be performed at approximately the same time of day. Subjects will be required to arrange for transportation home each day following completion of the experiments.

EEG RECORDING AND WORKING MEMORY TASK The EEG portion of this project will be conducted in the Neuroinformatics Lab in the J. Crayton Pruitt Family Department of Biomedical Engineering at the University of Florida. Subjects will be comfortably seated inside an acoustically and electrically shielded booth designed to reduce ambient noise and 60 Hz activity. 128 small electrodes will be placed on the research subjects' scalp using spandex electrode cap. Standard procedures are used to reduce the electrical resistance at each recording site by injecting a small amount of conductive gel into each electrode holder on the cap. The scalp in each electrode site will be rubbed lightly before the gel injected. In addition, seven additional flat-type electrodes are to be used, (a) two for each lateral side of both eyes, (b) two for the above and below of the left eye, (c) two for right behind each ear and (d) one for one of the arms depending on the subject's hand orientation.

The subject then is seated on a non-metal wooden chair in front of a computer screen inside the electromagnetically and acoustically shielded chamber located in the lab. The subject should memorize different set of numbers (maximum of five different digits) that will appear on the screen. A few seconds later a probe (one digit number) will appear on the screen and the subject need to responds as quickly as possible by pressing a button to indicate whether the number belongs to the set.

One hour paradigm consists of four 15 minute blocks. Practice block will be given before the actual one and one minute break time between the blocks will be given. Investigators can communicate with the subject either by looking at the closed-circuit TV (CCTV) system from outside or by talking through the wired radio system during the task.

NEUROPSYCHOLOGY BATTERY A battery of neuropsychological tests that includes measures from our cognitive AED protocol as well as additional language-specific measures will be used: Controlled Oral Word Association Test (COWA), which tests the ability to generate words beginning with a specific letter of the alphabet; Action Verb Fluency, in which the subject lists as many action verbs (run, climb) as they can in one minute; Category Fluency, in which the subject lists as many names (i.e., of animals, pieces of clothing, etc) as they can in one minute; Category Switching, where the subject switches between recall of names from two different categories, i.e., between fruits and furniture; Hopkins Verbal Learning Test (HVLT),which offers a brief assessment of verbal learning and memory (recognition and recall) for individuals 16 years and older. It is a word list learning task; Symbol Digit Modalities Test (SDMT), a test of graphomotor and psychomotor speed. Additional psychological tests that will be administered include Boston Naming Test, action verb fluency test, and the Boston Diagnostic Aphasia Examination Picture Description Task (PictA) in which the subject is asked to describe a black-and-white schematic pencil drawing of a scene containing several types of elicitation stimuli. (<5 min). Alternate versions of this task include the Minnesota Test for Differential Diagnosis of Aphasia (PictB) and the Nichols-Brookshire "Rescue" Picture Description Task (PictC) Administration of this battery will take approximately 20-25 minutes. All tests will be audiotaped for further speech and language analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women (post menopausal or using approved birth control methods

Exclusion Criteria:

* Presence of clinically significant cardiovascular, endocrine, hematopoietic, hepatic, neurologic, psychiatric, or renal disease
* Presence or history of drug or alcohol abuse
* The use of concomitant medications which are known to affect topiramate or the use of any concomitant medications that may alter cognitive function, including antidepressants, anxiolytics, psychostimulants such Ritalin, prescribed analgesics, and antipsychotics.
* Prior adverse reaction to or prior hypersensitivity to topiramate or to related compounds
* Subjects who have received any investigational drug within the previous thirty days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Controlled Oral Word Association test | 6 hours
  generative verbal fluency

IPD SHARING:
Plan to Share IPD: Undecided